CLINICAL TRIAL: NCT03135782
Title: Integrating Tobacco Cessation Coaching Sessions Into Radiation Medicine Treatment: A Pilot Study
Brief Title: Provider Training in Increasing Patient Tobacco Cessation Counseling and Referrals for Patients With Cancer Undergoing Radiation Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, John Holland, Associate Professor, OHSU Knight Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00016428; NCI-2017-00576 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00016428 (Other: OHSU Knight Cancer Institute)
Record Dates: First submitted 2017-04-26; First posted 2017-05-01 (Actual); Last update posted 2021-03-05 (Actual); Status verified 2021-03

CONDITIONS: Breast Carcinoma; Caregiver; Head and Neck Carcinoma; Lung Carcinoma; Prostate Carcinoma; Tobacco Use
MeSH Terms: conditions — Breast Neoplasms; Lung Neoplasms; Prostatic Neoplasms; Tobacco Use

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Health Services Research (Chart review, training, coaching) (Experimental): MEDICAL CHART REVIEW: Medical charts from patients with diagnoses of head and neck cancer, lung cancer, prostate cancer, or breast cancer are reviewed at months 1-12 to determine the frequency of tobacco assessments and documentation of discussions with patients regarding tobacco use and utilization of cessation resources as before and after the proposed training.
  PROVIDER TRAINING: Providers undergo training to use patient coaching such as the 5A's (Ask, Advise, Assess, Assist, and Arrange), to conduct regular tobacco intake assessment using motivational interviewing techniques. Providers also undergo training to use public/community tobacco cessation resources for patients ready to quit within six weeks, and have access to pharmacy residents for ad-hoc prescribing questions.
  PATIENT COACHING: Patients attend 4 phone or in-person motivational interviewing coaching sessions over 30-45 minutes for 6-8 weeks or longer as needed.
  Interventions: Other: Communication Skills Training; Other: Medical Chart Review; Other: Questionnaire Administration; Other: Tobacco Cessation Counseling

INTERVENTIONS:
Other: Communication Skills Training — Undergo motivational interviewing training
Other: Medical Chart Review — Undergo medical chart review
  Other Names: Chart Review
Other: Questionnaire Administration — Ancillary studies
Other: Tobacco Cessation Counseling — Attend phone or in-person motivational interviewing coaching sessions

SUMMARY:
This pilot clinical trial studies how well provider training works in increasing patient tobacco cessation counseling and referrals for patients with cancer undergoing radiation therapy. Health care provider training in motivational interviewing techniques and utilizing tobacco cessation resources may help doctors understand how health care providers can effectively increase their confidence in talking to patients about tobacco cessation counseling.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if training providers on tobacco cessation resources increases the frequency of counseling and referrals at initial and follow-up consultations for cancer patients who use tobacco and are scheduled to receive radiation at Oregon Health and Science University (OHSU).

SECONDARY OBJECTIVES:

I. Increase provider frequency of tobacco use quantification and type. II. Increase frequency of provider assessment of tobacco cessation readiness in current users.

III. Increase frequency and types of tobacco cessation resources and medicines offered and utilized.

IV. Increase frequency and type of follow-up planned if referred to cessation resource.

OUTLINE:

MEDICAL CHART REVIEW: Medical charts from patients with diagnoses of head and neck cancer, lung cancer, prostate cancer, or breast cancer are reviewed at months 1-12 to determine the frequency of tobacco assessments and documentation of discussions with patients regarding tobacco use and utilization of cessation resources as before and after the proposed training.

PROVIDER TRAINING: Providers undergo training to use patient coaching such as the 5A's (Ask, Advise, Assess, Assist, and Arrange), to conduct regular tobacco intake assessment using motivational interviewing techniques. Providers also undergo training to use public/community tobacco cessation resources for patients ready to quit within six weeks, and have access to pharmacy residents for ad-hoc prescribing questions.

PATIENT COACHING: Patients attend 4 phone or in-person motivational interviewing coaching sessions over 30-45 minutes for 6-8 weeks or longer as needed.

ELIGIBILITY:
Inclusion Criteria:

* MEDICAL CHART REVIEW
* Pre-intervention: 200 patient records between January 1, 2016 and December 31, 2016 are subject to review; the first 50 records with a diagnoses of each cancer type: head and neck, lung, prostate, or breast will be utilized for the review
* Post-intervention: 200 patient records receiving care beginning six months post training are subject to review; the first 50 records with a diagnoses of head and neck, lung, prostate, or breast will be utilized
* PROVIDER TRAINING
* OHSU Radiation Medicine department has agreed to participate as pilot department for this project; all active Radiation Medicine providers are requested to participate in the training; providers have the option to not participate
* TOBACCO CESSATION COACHING
* Patients who are at least 18 years of age
* Speak English
* Report tobacco use within the past 7 days
* Willing to consider quitting smoking
* Patients must be willing to meet four times in person or on the phone to discuss tobacco use
* Patients must be willing to be audio recorded during the sessions
* Patients who meet this criteria will be referred to OHSU Health Promotion Sports Medicine researcher, Carol DeFrancesco, to complete assessment using stages of change tobacco use readiness ruler and question set
* Patient smoking status will be documented in their electronic health record, per routine care

Exclusion Criteria:

* Vulnerable Populations

  * The following groups will be excluded from participation:

    * Children
    * Decisionally impaired adults
    * Prisoners
    * Pregnant women

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2020-09-23 (Actual); Study Completion 2020-09-23 (Actual)

PRIMARY OUTCOMES:
Change in frequency of tobacco counsel | Baseline up to 24 months
  Will be compared between the cohort of pre and post intervention. Will be summarized using descriptive statistics and compared using chi-square test by tumor type.

SECONDARY OUTCOMES:
Change in frequency and type of follow-up planned if referred to cessation resource assessed by medical chart review | Baseline up to 24 months
  Will be summarized using descriptive statistics and compared using chi-square test by tumor type.
Change in frequency and types of tobacco cessation resources and medicines offered and utilized assessed by medical chart review | Baseline up to 24 months
  Will be tested using a chi-squared test. If any expected cell count in the contingency table is lower than 5, we will instead use Fisher's exact test.
Change in frequency of provider assessment of tobacco cessation readiness in current users assessed by medical chart review | Baseline up to 24 months
  Will be summarized using descriptive statistics and compared using chi-square test by tumor type.
Change in provider frequency of tobacco use quantification and type assessed by medical chart review | Baseline up to 24 months
  Will be summarized using descriptive statistics and compared using chi-square test by tumor type. Will be tested using Z tests of proportion.

CONTACTS AND LOCATIONS:
Overall Officials: John Holland, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States

REFERENCES:
- [Background] Holland JM, Holland E, Chen Y, Brown SA. Smoking history and cessation discussions in cancer patients receiving definitive radiotherapy: Do we treat all patients equally? Tob Prev Cessat. 2020 May 22;6:31. doi: 10.18332/tpc/120308. eCollection 2020. PMID 32760866